CLINICAL TRIAL: NCT05057767
Title: Impact of Timing of Midazolam Administration on Incidence of Postoperative Nausea and Vomiting in Patients Undergoing Laparoscopic Gynecological Surgery; a Randomized Double-blinded Controlled Study
Brief Title: Impact of Timing of Midazolam Administration on Incidence of Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Samar Rafik Mohamed Amin, lecturer of anesthesia and surgical ICU, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC-12-8-2021
Record Dates: First submitted 2021-09-13; First posted 2021-09-27 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-induction Group (I) (Experimental): will receive intravenous midazolam premedication 2mg in a volume of 3 ml, 15 minutes before induction of anesthesia
  Interventions: Drug: Midazolam injection
- Pre-extubation Group (II) (Experimental): will receive intravenous midazolam 2mg in a volume of 3 ml 30 minutes before extubation at the end of surgery
  Interventions: Drug: Midazolam injection
- Control Group (III) (Placebo Comparator): will receive 3 ml normal saline 15 minutes before induction of anesthesia plus 3 ml normal saline 30 minutes before extubation at the end of surgery.
  Interventions: Drug: Midazolam injection

INTERVENTIONS:
Drug: Midazolam injection — No premedication will be given to Patients in the group undergoing a standardized anesthesia protocol which include induction with thiopental (5 mg/kg) and fentanyl (1-2 μg/kg). Atracurium will be used as a muscle relaxant. After tracheal intubation, anesthesia will be maintained with isoflurane in a concentration of 0.8%-1.2%. Ventilation will be adjusted to produce normocapnia. At the end of surgery, reversal of residual neuromuscular blockade will be accomplished using i.v. atropine 20 μg/Kg and neostigmine 40 μg/kg.

SUMMARY:
Postoperative nausea and vomiting (PONV), defined as nausea and/or vomiting occurring within 24 hours after surgery, affects between 20% and 30% of patients, As many as 70% to 80% of patients at high risk may be affected. The etiology of PONV is thought to be multifactorial, involving individual, anaesthetic and surgical risk factors. PONV results in increased patient discomfort and dissatisfaction and in increased costs related to length of hospital stay. Serious medical complications such as pulmonary aspiration, although uncommon, are also associated with vomiting.

Patients with a higher risk of PONV often require a combination or multimodal approach of 2 or more interventions for effective risk reduction. Thus, researchers have explored additional nontraditional antiemetics, such as midazolam, that would aid in the multimodal prevention of PONV.

DETAILED DESCRIPTION:
Midazolam is often administered in the perioperative period to reduce anxiety in addition to causing sedation and amnesia. The pharmacologic qualities allow for a rapid onset, short duration, and short half-life. The clinical effects of midazolam result from an agonist action on the γ-aminobutyric acid A (GABAA) receptor throughout the central nervous system. Benzodiazepines do not work directly on the GABA receptor, so there is a physiologic ceiling effect, which contributes to their safety and low toxicity.

Although the exact antiemetic mechanisms remain unknown, researchers postulate that midazolam works on the chemoreceptor trigger zone by reducing the synthesis, release, and postsynaptic dopamine. It remains debatable whether midazolam reduces dopamine directly or blocks the reuptake of adenosine leading to an adenosine-mediated reduction of dopamine release. Additionally, the binding of midazolam to the GABA benzodiazepine complex may cause dopaminergic neuronal activity and the release of 5-hydroxytryptamine. The reduction of PONV may also be a secondary effect of the anxiolytic properties of benzodiazepines.

Despite literature demonstrating the PONV benefits of midazolam in the perioperative period, But the timing of administration of this drug is still not well established. As it is known that it has half-life of about 1.5 - 2.5 hours and the controversies remain whether to administer this drug preoperatively or postoperatively to prevent PONV. So this comparative study is designed to know the better time for administration of this drug to prevent PONV and to improve patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* aged twenty to sixty years old
* The American Society of Anesthesiologists (ASA) physical status classification grade I or II
* Scheduled for laparoscopic gynecological surgeries under general anesthesia.

Exclusion Criteria:

* Patients who have gastrointestinal disorders,
* histories of PONV after a previous surgery,
* Renal or liver dysfunction,
* history of motion sickness,
* Have received any opioid, steroid, or antiemetic medication in the 24hs before surgery, and
* Pregnant or menstruating women.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Post Operative Nausea Vomiting assessment | 24 hours postoperative
  Nausea will be recorded according to the following scale: 0 none; 1 mild (patient able to eat); 2 moderate (oral intake significantly decreased); and 3 severe (no significant oral intake necessitating iv fluid). The absence of nausea will be defined as complete protection from nausea. An emetic episode will be defined as a single vomit or retch, or any number of continuous vomiting episodes or retches (one emetic episode should be separated from another by an absence of vomiting or retching for at least 1 min). The absence of emetic episodes will be defined as complete protection from vomiting.

SECONDARY OUTCOMES:
requirements of rescue antiemetic | 24 hours postoperative
  Rescue medication (metoclopramide 10 mg) will be given intravenously if patient is nauseous for more than 15 min or experiences retching or vomiting during the observation periods. The treatment will be repeated if necessary
Observer's Assessment of Alertness/ Sedation (OAA/S) scale | 120 minutes postoperative
  a six-point scale ranging from 5 to 0 that involves eliciting a response to increasingly intense stimuli that begin with speaking with a normal voice to prodding or shaking and finally to a painful stimulus (trapezius squeeze).
Pain intensity score | 24 hours postoperative
  measured with a visual analog scale (VAS) from 0 (no pain) to 10 (the worst possible pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Rafik Mohamed Amin, Banhā, Qalyubia Governorate, Egypt